CLINICAL TRIAL: NCT05825209
Title: Food-Grown Magnesium Supplement on Sleep Quality/Quantity in a Healthy Adult Population: A Double Blind Randomized Placebo-controlled Study
Brief Title: Effectiveness of Food-grown Magnesium on Sleep Quality/Quantity
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: RDC Clinical Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MAGSLE
Record Dates: First submitted 2023-03-27; First posted 2023-04-24 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-03

CONDITIONS: Sleep
MeSH Terms: interventions — microcrystalline cellulose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Food-Grown Magnesium (Active Comparator): Food-grown magnesium in capsule form - taken as 2 capsules, orally with water 1 hour before sleep.
  Interventions: Drug: Food-Grown Magnesium
- Microcrystalline cellulose (Placebo Comparator): Microcrystalline cellulose in capsule form - taken as 2 capsules, orally with water 1 hour before sleep.
  Interventions: Drug: Microcrystalline cellulose

INTERVENTIONS:
Drug: Food-Grown Magnesium — 1 daily dose of 2 capsules equivalent to 80mg food-grown magnesium (40mg per capsule)
  Arms: Food-Grown Magnesium
Drug: Microcrystalline cellulose — 1 daily dose of 2 capsules containing microcrystalline cellulose
  Arms: Microcrystalline cellulose

SUMMARY:
This is a double-blind randomised placebo-controlled trial to evaluate orally-dosed food-grown magnesium compared to placebo on improvement in sleep quality and quantity as well as quality of life in otherwise healthy participants aged 18 years and older.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years or older
* Otherwise healthy
* Disturbed sleeping pattern (defined as difficulty falling asleep, waking up during the sleep cycle or waking up too early and being unable to fall back to sleep)
* Able to provide informed consent
* Agree not to change current diet/exercise or not to use other medicines or supplements for sleep or anxiety other than the test product during entire study period.
* Agree not to participate in another clinical trial while enrolled in this trial

Exclusion Criteria:

* Unstable or serious illness (e.g. serious mood disorders such as depression or bipolar disorder, neurological disorders such as MS, kidney disease, liver disease, GIT conditions, heart conditions, diabetes, thyroid gland function) (1)
* History of renal function impairment
* Regular sleeping pattern
* Current malignancy (excluding BCC) or chemotherapy or radiotherapy treatment for malignancy within the previous 2 years
* Receiving/prescribed coumadin (Warfarin), heparin, dalteparin, enoxaparin or other anticoagulation therapy
* Receiving/prescribed sleep or anxiety medication/aid
* Sleep apnea
* Diagnosed or consistent gastrointestinal issues that disrupt sleep
* Active smokers, nicotine use, drug abuse
* Chronic past and/or current alcohol use (>14 alcoholic drinks week)
* Allergic to any of the ingredients in active or placebo formula
* People with serious mood disorders (such as depression, anxiety and bipolar disorder) will be excluded
* Those suffering from insomnia or have night-shift employment and unable to have a normal night's sleep (2)
* People suffering any neurological disorders such as MS
* Pregnant or lactating woman
* Any condition which in the opinion of the investigator makes the participant unsuitable for inclusion
* Participants who have participated in any other clinical trial during the past 6 months
* Clinically significant acute or chronic inflammation, or connective tissue disease or arthritis
* History of infection in the month prior to the study
* Regularly taking stimulants (e.g., coffee, caffeine supplements, caffeine containing beverages) 2 hours before bed
* Disturbed sleeping pattern caused by external factors (e.g., children, partner, noises)

  1. An unstable illness is any illness that is currently not being treated with a stable dose of medication or is fluctuating in severity. A serious illness is a condition that carries a risk of mortality, negatively impacts quality of life and daily function and/or is burdensome in symptoms and/or treatments.
  2. Insomnia has been excluded as it is a significant health condition, and we are testing on otherwise healthy participants (as per TGA complementary medicine requirements)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2023-04-06 (Actual); Primary Completion 2023-07-04 (Actual); Study Completion 2023-07-04 (Actual)

PRIMARY OUTCOMES:
Change in sleep quality by self-reported assessment via Consensus Sleep Diary - Morning Administration (CSD-M). | Baseline, week 1, week 4 and week 8
  Change in sleep quality by self-reported assessment via Consensus Sleep Diary - Morning Administration (CSD-M). Sleep quality is assessed by a 5 category rating from 'Very poor' to 'Very good'. Sleep quality is also assessed by a 5 category rating of the degree of rested state from 'Not at all rested' to "Very well-rested'
Change in sleep quantity by self-reported assessment via Consensus Sleep Diary - Morning Administration (CSD-M). | Baseline, week 1, week 4 and week 8
  Change in sleep quantity, as defined as the collective amount of sleep obtained in a given period, by self-reported assessment via Consensus Sleep Diary - Morning Administration (CSD-M).

SECONDARY OUTCOMES:
Change in quality of life | Baseline and week 8
  Change in quality of life as assessed by the Short Form 36 Health Survey Questionnaire (SF36) which consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability.
Change in height in anthropometry measurements | Baseline and week 8
  Height as measured by stadiometer in centimeters
Change in weight in anthropometry measurements | Baseline and week 8
  Weight as measured by digital scales in kilograms
Change in BMI in anthropometry measurements | Baseline and week 8
  Height and will be combined to report BMI in kg/m2
Change in sleep onset time as assessed by the Pittsburgh Sleep Quality Index (PSQI) | Baseline, week 4 and week 8
  Change in sleep onset time as assessed by the Pittsburgh Sleep Quality Index (PSQI). Seven component scores are derived, each scored 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality.
Change in sleep onset time as assessed by self-reported assessment of sleep quality via Consensus Sleep Diary - Morning Administration (CSD-M). | Baseline, week 1, week 4 and week 8
  Change in sleep onset time as assessed by self-reported assessment of sleep quality via Consensus Sleep Diary - Morning Administration (CSD-M). Participants are asked "How long did it take you to fall asleep?"
Change in sleep onset time as assessed by wrist actigraphy | Baseline, week 1, week 4 and week 8
  Change in sleep onset time as assessed by wrist actigraphy which measures wrist movements to assess sleep or waking state.
Change in sleep pattern disturbance as assessed by the Pittsburgh Sleep Quality Index (PSQI) | Baseline, week 4 and week 8.
  Change in sleep pattern disturbance as assessed by the Pittsburgh Sleep Quality Index (PSQI). Seven component scores are derived, each scored 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality.
Change in sleep pattern disturbance as assessed by wrist actigraphy | Baseline, week 1, week 4 and week 8
  Change in sleep pattern disturbance as assessed by wrist actigraphy which measures wrist movements to assess sleep or waking state.
Change in daytime sleepiness as assessed by the Epworth Sleepiness Scale (ESS) | Baseline, week 4 and week 8
  Change in daytime sleepiness as assessed by the Epworth Sleepiness Scale (ESS) which is a list of eight situations in which you rate your tendency to become sleepy on a scale of 0, no chance of dozing, to 3, high chance of dozing. The ESS score (the sum of 8 item scores) can range from 0 to 24. The higher the ESS score, the higher that person's average sleep propensity or their 'daytime sleepiness'.
Change in restless legs symptoms as assessed by the Restless Legs Syndrome Questionnaire | Baseline, week 4 and week 8
  Change in restless legs symptoms as assessed by the Restless Legs Syndrome Questionnaire. Ten component scores are derived, each scored 0 (none) to 4 (very severe). The component scores are summed to produce a global score (range 0 to 40). Higher scores indicate more severe symptoms.
Change in anxiety and stress levels as assessed by the Depression Anxiety and Stress Scale (DASS-21) | Baseline and week 8
  Change in anxiety and stress levels as assessed by the Depression Anxiety and Stress Scale (DASS-21) comprising 21 questions all with a rating scale from 0 (Did not apply to me at all) to 3 (Applied to me very much or most of the time). The total score represents overall distress (0 to 30), with higher scores indicating more severe distress or a greater number of symptoms.

OTHER OUTCOMES:
Adverse Events self-reported by participants | 8 week period from enrolment to participant conclusion
  Adverse Events self-reported by participants
Change in medication use | Baseline, week 1, week 4 and week 8
  Change in medication use self-reported by participants
Investigational product dosing compliance | Baseline, week 1, week 4 and week 8
  Investigational product dosing compliance self-reported by participants

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Rao, PhD, Principal Investigator — RDC Clinical Pty Ltd
Locations (1):
- RDC Global Pty Ltd, Brisbane, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared